CLINICAL TRIAL: NCT00002257
Title: A Randomized Controlled Study of the Efficacy and Safety of Maintenance Treatment With Oral Ganciclovir for Newly Diagnosed Cytomegalovirus Retinitis in People With AIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 059B; ICM 1653
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1992-07

CONDITIONS: Cytomegalovirus Retinitis; HIV Infections
Keywords: Retinitis; Ganciclovir; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Cytomegalovirus Retinitis; HIV Infections; Retinitis; Multiple Acyl Coenzyme A Dehydrogenase Deficiency; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome | interventions — Ganciclovir

INTERVENTIONS:
Drug: Ganciclovir

SUMMARY:
To compare the time to progression of CMV retinitis between oral ganciclovir and IV ganciclovir during 20 weeks of maintenance treatment. To compare the safety and tolerance of oral ganciclovir with IV ganciclovir therapy during 20 weeks of maintenance treatment. To describe the safety and tolerance of oral ganciclovir treatment when given concurrently with anti-retroviral treatment, e.g. zidovudine or ddI. To describe the survival of people with AIDS and CMV retinitis.

DETAILED DESCRIPTION:
Approximately 150 subjects with AIDS and newly diagnosed CMV retinitis will be enrolled in the study to achieve 120 randomized subjects. Eligible subjects will have CMV retinitis which has been diagnosed within one month of study entry by an ophthalmologist using indirect ophthalmoscopy. Subjects will be accrued by recruitment or referral. Anyone who volunteers for the study, meets the eligibility criteria, and signs an informed consent will be eligible for entry.

ELIGIBILITY:
Inclusion Criteria

Patients must have the following:

* Confirmation of HIV infection by HIV-antibody testing, p24 antigen assay, or culture of HIV, or have diagnosis of AIDS by CDC criteria.
* CMV retinitis diagnosed within one month of study entry.
* Understand the nature of the study, agree to its provisions, and sign the informed consent approved by the appropriate institutional review board and Syntex.

Exclusion Criteria

Concurrent Medication:

The following are excluded:

* Antimetabolites. Alkylating agents. Selected nucleoside analogs. Selected Cytokines.

Patients with the following are excluded:

* Persistent diarrhea, nausea, or abdominal pain or other clinically significant GI symptoms or uncontrolled gastrointestinal disease. Diarrhea is defined as 3 or more unformed stools per day.
* Have ocular media opacities (corneal, lenticular, or vitreal) preventing ophthalmologic retinal assessment and photography.
* Have ocular conditions requiring immediate surgical correction (e.g. retinal tear or detachment).
* Require continuation of concomitant medications precluded by this protocol, e.g., antimetabolites, alkylating agents, selected nucleoside analogs, and selected cytokines and other medications listed in the protocol.
* History of hypersensitivity to acyclovir or ganciclovir.
* Dementia, decreased mentation or other encephalopathic signs and symptoms which would interfere with the ability of the subject to give informed consent or comply with the protocol.

Prior Medication:

The following are excluded:

- Previous use of anti-cytomegalovirus drug (e.g., ganciclovir, foscarnet, FIAC, or CMV hyperimmune globulin) within one month of study entry.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150

CONTACTS AND LOCATIONS:
Locations (13):
- United States (12):
  - East Bay AIDS Ctr, Berkeley, California
  - Davies Med Ctr / c/o HIV Institute, San Francisco, California
  - Dr David Busch, San Francisco, California
  - Georgetown Univ Med Ctr, Washington D.C., District of Columbia
  - Med Service, Miami, Florida
  - Miami Veterans Administration Med Ctr, Miami, Florida
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Beth Israel Deaconess Med Ctr, Boston, Massachusetts
  - New York Univ Med Ctr, New York, New York
  - Cornell Univ Med College, New York, New York
  - Buckley Braffman Stern Med Associates, Philadelphia, Pennsylvania
  - Univ TX Galveston Med Branch, Galveston, Texas
- Saint Paul's Hosp, Vancouver, British Columbia, Canada